CLINICAL TRIAL: NCT03112655
Title: Diagnostic Tools for Human African Trypanosomiasis Elimination and Clinical Trials: WP4 Early Test-of-cure
Brief Title: Diagnostic Tools for Human African Trypanosomiasis Elimination and Clinical Trials: Early Test-of-cure
Acronym: DiTECT-WP4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Institute of Tropical Medicine, Belgium (Other); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Ministry of Public Health, Democratic Republic of the Congo (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: DiTECT-HAT-WP4
Record Dates: First submitted 2017-03-31; First posted 2017-04-13 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-01

CONDITIONS: African Trypanosomiasis; African; Trypanosomiasis, West; Sleeping Sickness; West African; Trypanosoma Brucei Gambiense; Infection
Keywords: diagnosis; sensitivity; specificity; therapeutic outcome; cerebrospinal fluid
MeSH Terms: conditions — Trypanosomiasis, African; Trypanosomiasis; Infections; Disease; Hypersensitivity

STUDY DESIGN:
Masking Description: The reference laboratory, generating the results for the index test, is masked for results obtained at the clinical trial site (determining the standard reference).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human african trypanosomiasis patient (Experimental): RNA, neopterin and 5-hydroxytryptophan detection
  Interventions: Diagnostic Test: RNA and neopterin detection

INTERVENTIONS:
Diagnostic Test: RNA and neopterin detection — Detection of spliced leader RNA will be performed on blood and cerebrospinal fluid taken before treatment, 11 days after treatment, 6, 12 and 18 months after treatment. Neopterin and 5-hydroxytryptophan will be quantified in cerebrospinal fluid taken at the same time points.
  Other Names: Reverse transcriptase real-time PCR Trypanozoon SL-RNA; Neopterin & 5-hydroxytryptophan EIA, Mybiosource

SUMMARY:
The study validates the diagnostic performance of cerebrospinal fluid neopterin quantification and of blood and cerebrospinal fluid trypanosomal spliced leader RNA detection for assessing outcome after treatment of human African trypanosomiasis.

DETAILED DESCRIPTION:
In the last decade, the prevalence of Trypanosoma brucei gambiense human African trypanosomiasis (HAT) has fallen and HAT has been targeted for elimination. Development of safe and efficacious drugs for HAT, applicable in an elimination context, is considered as a high priority. The drug developmental process is however slowed down by the need to follow-up treated patients for 18 months to decide on cure. For timely diagnosis of treatment failure in clinical trials, patients should have control visits with follow-up examinations at 6, 12 and 18 months after treatment. Furthermore, due to repeated lumbar punctures, treated patients refrain to present for control visits spontaneously, and tend not to comply with follow-up. Clinical trials on new drugs for HAT would therefore be accelerated by availability of an early test of cure. Trypanosomal spliced leader (SL)-RNA, neopterin & 5-hydroxytryptophan are good candidates for accurate and shortened treatment follow-up. In particular SL-RNA detection in blood offers an opportunity for non-invasive post-treatment follow-up.

The objective of the DiTECT-HAT-WP4 study is to validate the diagnostic performance of cerebrospinal fluid neopterin & 5-hydroxytryptophan quantification and of blood and cerebrospinal fluid trypanosomal spliced leader RNA detection for assessing treatment outcome. The DiTECT-HAT-WP4 study is embedded into an ongoing therapeutic phase II/III study (DNDi-OXA-02-HAT) testing a new oral single dose drug against HAT. Within the Framework of the therapeutical trial, patients will have post-treatment examinations, including blood and cerebrospinal fluid examination at day 11, and during follow-up at month 6, month 12 and month 18. Combination of DiTECT-HAT-WP4 with this ongoing clinical trial allows evaluation of new treatment outcome assessment markers during follow-up without the need for additional lumbar or venipunctures. The volumes of venous blood and cerebrospinal fluid taken will be increased by 2.5 mls for the DiTECT-HAT-WP4 study.

Reverse transcriptase real time PCR for spliced leader RNA detection in blood and cerebrospinal fluid and neopterin detection will be carried out in the reference laboratory in Kinshasa, (index tests). The reference laboratory will be blinded to the results of the reference standard. For evaluation of diagnostic performance of the index tests, the reference standard will consist of classification of treatment outcome according to international standards applied for the clinical trial. Receiver operator curves, sensitivity and specificity of the different index tests for treatment outcome assessment will be determined at each follow-up time point. If sufficiently accurate, trypanosomal spliced leader RNA detection in blood would allow post-treatment follow-up without the need for lumbar punctures. Improved treatment outcome assessment will not only facilitate follow-up by avoiding the feared lumbar puncture but also speed up the development and implementation of new drugs. In addition, it will also improve management of patients in routine. The proposed research will impact on clinical decision and treatment outcomes, and contribute to successful HAT elimination.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for participation in DNDi-OXA-02-HAT clinical trial

Exclusion Criteria:

* Excluded for DNDi-OXA-02-HAT clinical trial; No informed consent for participation in the DiTECT-HAT-WP4 study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of SL-RNA detection in blood, SL-RNA detection in cerebrospinal fluid and of neopterin & 5-hydroxytryptophan quantification in cerebrospinal fluid for relapse after human African trypanosomiasis treatment | 18 months
  Index tests: qualitative detection of SL-RNA in blood, qualitative detection of SL-RNA in cerebrospinal fluid, neopterin & 5-hydroxytryptophan quantification in cerebrospinal fluid.
  Reference standard: classification according to the WHO 2015 criteria as relapse or probable relapse within 18 months after treatment for human African trypanosomiasis
Specificity of SL-RNA detection in blood, SL-RNA detection in cerebrospinal fluid and of neopterin & 5-hydroxytryptophan quantification in cerebrospinal fluid for cure after human African trypanosomiasis treatment | 18 months
  Index tests: qualitative detection of SL-RNA in blood, qualitative detection of SL-RNA in cerebrospinal fluid, neopterin & 5-hydroxytryptophan quantification in cerebrospinal fluid.
  Reference standard: classification according to the WHO 2015 criteria as cure or probable cure 18 months after treatment

SECONDARY OUTCOMES:
Sensitivity and specificity SL-RNA detection in blood for outcome assesment after treatment for human African trypanosomiasis | post treatment day 11, month 6, month 12 and month 18
  Index tests: qualitative detection of SL-RNA in blood post treatment day 11, month 6, month 12 and month 18.
  Reference standard: Human African trypanosomiasis treatment outcome classification according to the WHO 2015 criteria
Sensitivity and specificity SL-RNA detection in cerebrospinal fluid for outcome assesment after treatment for human African trypanosomiasis | post treatment day 11, month 6, month 12 and month 18
  Index tests: qualitative detection of SL-RNA in cerebrospinal fluid at post treatment day 11, month 6, month 12 and month 18.
  Reference standard: Human African trypanosomiasis treatment outcome classification according to the WHO 2015 criteria
Sensitivity and specificity by ROC analysis of neopterin & 5-hydroxytryptophan quantification in cerebrospinal fluid for outcome assesment after treatment for human African trypanosomiasis | post treatment day 11, month 6, month 12 and month 18
  Index tests: quantitative detection of neopterin & 5-hydroxytryptophan in cerebrospinal fluid at post treatment day 11, month 6, month 12 and month 18.
  Reference standard: Human African trypanosomiasis treatment outcome classification according to the WHO 2015 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Lejon, PhD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (1):
- Programme Nationale de Lutte contre la trypanosomiase humaine Africaine, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez-Andrade P, Camara M, Ilboudo H, Bucheton B, Jamonneau V, Deborggraeve S. Diagnosis of trypanosomatid infections: targeting the spliced leader RNA. J Mol Diagn. 2014 Jul;16(4):400-4. doi: 10.1016/j.jmoldx.2014.02.006. Epub 2014 May 9. PMID 24814957
- [Background] Ilboudo H, Camara O, Ravel S, Bucheton B, Lejon V, Camara M, Kabore J, Jamonneau V, Deborggraeve S. Trypanosoma brucei gambiense Spliced Leader RNA Is a More Specific Marker for Cure of Human African Trypanosomiasis Than T. b. gambiense DNA. J Infect Dis. 2015 Dec 15;212(12):1996-8. doi: 10.1093/infdis/jiv337. Epub 2015 Jun 16. PMID 26080371
- [Background] Tiberti N, Lejon V, Hainard A, Courtioux B, Robin X, Turck N, Kristensson K, Matovu E, Enyaru JC, Mumba Ngoyi D, Krishna S, Bisser S, Ndung'u JM, Buscher P, Sanchez JC. Neopterin is a cerebrospinal fluid marker for treatment outcome evaluation in patients affected by Trypanosoma brucei gambiense sleeping sickness. PLoS Negl Trop Dis. 2013;7(2):e2088. doi: 10.1371/journal.pntd.0002088. Epub 2013 Feb 28. PMID 23469311
- [Background] Vincent IM, Daly R, Courtioux B, Cattanach AM, Bieler S, Ndung'u JM, Bisser S, Barrett MP. Metabolomics Identifies Multiple Candidate Biomarkers to Diagnose and Stage Human African Trypanosomiasis. PLoS Negl Trop Dis. 2016 Dec 12;10(12):e0005140. doi: 10.1371/journal.pntd.0005140. eCollection 2016 Dec. PMID 27941966
- [Derived] Ngay Lukusa I, Van Reet N, Mumba Ngoyi D, Mwamba Miaka E, Masumu J, Patient Pyana P, Mutombo W, Ngolo D, Kobo V, Akwaso F, Ilunga M, Kaninda L, Mutanda S, Mpoyi Muamba D, Valverde Mordt O, Tarral A, Rembry S, Buscher P, Lejon V. Trypanosome spliced leader RNA for diagnosis of acoziborole treatment outcome in gambiense human African trypanosomiasis: A longitudinal follow-up study. EBioMedicine. 2022 Dec;86:104376. doi: 10.1016/j.ebiom.2022.104376. Epub 2022 Nov 24. PMID 36436279
- [Derived] Ngay Lukusa I, Van Reet N, Mumba Ngoyi D, Miaka EM, Masumu J, Patient Pyana P, Mutombo W, Ngolo D, Kobo V, Akwaso F, Ilunga M, Kaninda L, Mutanda S, Muamba DM, Valverde Mordt O, Tarral A, Rembry S, Buscher P, Lejon V. Trypanosome SL-RNA detection in blood and cerebrospinal fluid to demonstrate active gambiense human African trypanosomiasis infection. PLoS Negl Trop Dis. 2021 Sep 17;15(9):e0009739. doi: 10.1371/journal.pntd.0009739. eCollection 2021 Sep. PMID 34534223
- See also: Human African trypanosomiasis: update of the methodological framework for clinical trials — http://apps.who.int/iris/bitstream/10665/173583/1/9789241508834_eng.pdf?ua=1
- See also: phase 1 study of drug now in phase 2/3 — https://clinicaltrials.gov/ct2/show/NCT01533961